CLINICAL TRIAL: NCT00550056
Title: Talking About Traumatic Events - A Randomized Controlled Dissemination Study of the Treatment of PTSD in an African Refugee Settlement
Brief Title: Treatment of Posttraumatic Stress Disorder by Trained Lay Counsellors in an African Refugee Settlement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: German Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NeEl-Ug-01
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Last update posted 2007-10-26 (Estimated); Status verified 2007-10

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD, Posttraumatic Stress Disorder, refugees, war
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): NET
  Interventions: Behavioral: Narrative Exposure Therapy
- 2 (Experimental): TC
  Interventions: Behavioral: Trauma Counselling
- 3 (No Intervention): Monitoring Group

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — Six session of Narrative Exposure Therapy
  Arms: 1
Behavioral: Trauma Counselling — Six sessions of Trauma Counselling, using a variety of skills incl. exposure methods following the skills of the therapist
  Arms: 2

SUMMARY:
The study is a pragmatic trial to study the efficacy of two active methods of psychotherapy for the treatment of posttraumatic stress disorder in a refugee camp in Africa. Treatment was administered by lay counsellors.

DETAILED DESCRIPTION:
Traumatic stress due to conflict and war causes major mental health problems in many resource-poor countries, especially those coping with displaced populations. There is a lack of intervention research in these populations.

Te purpose of this study was to examine whether trained lay counsellors can carry out effective treatment of PTSD in a refugee settlement.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of posttraumatic stress disorder

Exclusion Criteria:

* Drug abuse
* Psychosis
* Mental retardation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2003-01; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Symptoms measured with the Posttraumatic Diagnostic Scale | 9 months

SECONDARY OUTCOMES:
Expert diagnosis of PTSD established with CIDI interview | 9 months
Physical health symptoms assessed with a checklist | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Elbert, PhD, Principal Investigator — University of Konstanz
Locations (1):
- Nakivale Refugee Camp, Mbarara, Mbarara, Uganda